CLINICAL TRIAL: NCT07054593
Title: An Open-Label, Pilot Study Designed To Evaluate The Effect Of A Proton Pump Inhibitor On The Regional Composition Of The Gut Microbiota And Metabolic Profiles Of Health Volunteers Using The Capscan® Samplng Capsule
Brief Title: Effect of Proton Pump Inhibitors on Gut Microbiota Composition and Metabolites in Healthy Subjects Using CapScan
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Envivo Bio Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EB02
Record Dates: First submitted 2025-06-20; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CapScan — Gut sampling capsule

SUMMARY:
This study is designed to evaluate the effect of proton pump inhibitors on the regional composition of the gut microbiota and metabolic profiles of health volunteers using the CapScan collection capsule.

DETAILED DESCRIPTION:
Prospective, open-label, single-arm, non-randomized, single-center study designed to evaluate the effect of proton pump inhibitors on the regional composition of the gut microbiota and metabolic profiles of health volunteers using the CapScan collection capsule.

ELIGIBILITY:
INCLUSION CRITERIA

Subjects must meet all of the following criteria to be included in the study:

* Males or females 18 years of age or older and 85 years of age or younger at the time of the first Screening Visit.
* ASA Classification 1 or 2.
* For women of childbearing potential, negative urine pregnancy test within 7 days of Screening Visit. Willingness to use highly effective contraception during the entire study period (e.g.: implants, injectables, oral contraceptives, intra-uterine device or declared abstinence).
* Subject is fluent in English and understands the study protocol and informed consent and is willing and able to comply with study requirements and sign the informed consent form.

EXCLUSION CRITERIA

Subjects with any of the following conditions or characteristics must be excluded from the study:

* History of any of the following:

  * prior gastric or esophageal surgery, including bariatric surgery
  * bowel obstruction
  * gastric outlet obstruction
  * gastroparesis
  * acute diverticulitis
  * inflammatory bowel disease
  * ileostomy or colostomy
  * gastric or esophageal cancer
  * achalasia
  * active dysphagia or odynophagia
* Daily PPI use in the last 30 days
* Pregnancy or planned pregnancy within 30 days from Screening Visit, or breast-feeding
* Any form of active substance abuse or dependence (including drug or alcohol abuse), unstable medical or psychiatric disorder, or any chronic condition susceptible, in the opinion of the investigator, to interfere with the conduct of the study
* A clinical condition that, in the judgment of the investigator, could potentially pose a health risk to the subject while involved in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Identification of the gut microbial taxa using DNA sequencing of the samples obtained from the CapScan devices | 2 months
  A primary endpoint is to identify and quantitate the relative abundance of the gut microbial taxa using at least 3 million metagenomic DNA sequencing reads in at least 75% of the samples obtained from the CapScan devices.
Identification of the gut metabolites using liquid chromatography - mass spectrometry of the samples obtained from the CapScan devices | 2 months
  A primary endpoint is to identify at least 1,500 annotated gut metabolites from the intestinal tract in at least 75% of the samples obtained from the CapScan devices.

SECONDARY OUTCOMES:
Detect changes in composition of gut microbial taxa using DNA sequencing in subjects before and after omeprazole treatment | 2 months
  Evaluate the diversity, centroids and distributions of microbial taxa from sequenced CapScan samples of the study population from before and after omeprazole treatment.
Detect changes in composition of gut metabolites using liquid chromatography - mass spectrometry in subjects before and after omeprazole treatment | 2 months
  Evaluate the diversity, centroids and distributions of gut metabolites in CapScan samples of the study population from before and after omeprazole treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Silicon Valley Gastroenterology, Mountain View, California, United States